CLINICAL TRIAL: NCT00360984
Title: Can Hypoglycaemia Awareness Be Restored in Individuals With Type 1 Diabetes and Severe Hypoglycaemia Employing Optimised Subcutaneous Insulin Regime or Continuous Subcutaneous Insulin Infusion Pump
Brief Title: Prevention of Severe Hypoglycemia in Type 1 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Newcastle University (Other)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other); Newcastle Primary Care Trust (Other); Sanofi (Industry); Medtronic (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4044
Record Dates: First submitted 2006-08-04; First posted 2006-08-07 (Estimated); Last update posted 2006-08-07 (Estimated); Status verified 2006-07

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: CSII; insulin analog; severe hypoglycaemia; altered hypoglycaemia awareness; diabetes quality of life; CGMS
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Insulin Glargine

INTERVENTIONS:
Drug: insulin glargine
Device: continuous subcutaneous insulin infusion

SUMMARY:
Severe hypoglycaemia leading to collapse without warning is one of the most-feared complications for those with Type 1 diabetes. The aim of this study is to determine whether detection and targeted prevention of hypoglycaemia by using either an optimised subcutaneous insulin regime or continuous insulin regime can restore hypoglycaemia awareness in Type 1 diabetes. Following a 6-day continuous subcutaneous monitor glucose profile, participants will be randomised to 1 of 3 interventions: rigorous avoidance of hypoglycaemia on current insulin regime; targeted optimisation of subcutaneous insulin regime to avoid hypoglycaemia; or continuous subcutaneous insulin infusion. Symptomatic experience and severity of hypoglycaemia, pattern of hypoglycaemia on glucose profiling and, in selected individuals, response to hyperinsulinaemic hypoglycaemic clamp, will be compared over a 6 month period. It is envisaged that successful prevention of hypoglycaemia by one or more interventions may reverse altered hypoglycaemia awareness and prevent further episodes of severe hypoglycaemia.

DETAILED DESCRIPTION:
The unifying objective of the proposed unblinded randomized prospective study is to determine whether hypoglycaemia awareness in Type 1 diabetes can be restored by rigorous avoidance of hypoglycaemia addressed by one of the following interventions:

1. A non-targeted approach whereby pre-prandial glycaemic targets are raised from 4.5-7mmol/L to 7.2-8.3mmol/L and hypoglycaemia is rigorously avoided without specific alterations in subcutaneous insulin regime5
2. Optimisation of subcutaneous insulin regime employing pre-prandial short-acting insulin analogue in combination with once daily insulin Glargine targeted to prevent periods of hypoglycaemia identified by 24 hour glucose profiles
3. Insulin delivery by external pump (continuous subcutaneous insulin infusion) targeted to prevent periods of hypoglycaemia identified by 24 hour glucose profiles

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes
* recurrent severe hypoglycemia within the preceding 6 months
* attending the Newcastle Diabetes Centre

Exclusion Criteria:

* previous use of rapid- and long-acting insulin analogs used in an multiple daily insulin injection regimen
* previous use of continuous subcutaneous insulin infusion pump
* alcohol or drug abuse
* seizures unrelated to hypoglycemia.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21
Dates: Start 2003-05; Study Completion 2004-09

PRIMARY OUTCOMES:
prevention of severe hypoglycemia

SECONDARY OUTCOMES:
incidence of mild symptomatic hypoglycemia
HbA1C
Continuous Subcutaneous Glucose Monitoring System profiles
Altered Hypoglycemia Awareness survey
Hypoglycemia Fear Survey
Diabetes Quality Of Life of questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: James AM Shaw, MD; PhD, Principal Investigator — Newcastle University
Locations (1):
- Newcastle Diabetes Centre, Newcastle, Tyne and Wear, United Kingdom